CLINICAL TRIAL: NCT03418558
Title: Open-label, Phase II Study of Trastuzumab Emtansine in Patients With HER2-positive Metastatic Colorectal Cancer Progressing After Trastuzumab and Lapatinib: HERACLES RESCUE. (HER2 Amplification for Colo-rectaL Cancer Enhanced Stratification - REchallenge With her2 Selective Cytotoxic Uptake of Emtansine)
Brief Title: Study of Trastuzumab-emtansine in Patients With HER2-positive Metastatic Colorectal Cancer Progressing After Trastuzumab and Lapatinib.
Acronym: RESCUE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 011-IRCC-10IIS-15
Record Dates: First submitted 2018-01-24; First posted 2018-02-01 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: HER2 AMPLIFICATION
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HERACLES RESCUE (Experimental): Patients will receive trastuzumab-emtansine, iv 3,6 mg/kg every 21 days. Patients will receive study medication until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever come first
  Interventions: Drug: Trastuzumab emtansine

INTERVENTIONS:
Drug: Trastuzumab emtansine

SUMMARY:
This is a phase II, open label, multicenter study. Patients with advanced colon rectal cancer (CRC) harboring an amplified HER2 that have been previously treated and progressed with an aNti-HER2 treatment, will be treated with the anti HER2 antibody conjugate trastuzumab emtansine (TDM1).

Patients will receive study medication until disease progression, unacceptable toxicity, withdrawal of consent or death. Main objective of the study is the evaluation of objective response rate according to RECIST 1.1 criteria. Disease control rate, defined as the sum of complete, partial and stable disease patients over total patient, followed by response duration, time to progression and safety are secondary endpoints.

DETAILED DESCRIPTION:
In metastatic colorectal cancer, HER2 amplified patients relapsing after initial long-lasting response to the anti HER combination of trastuzumab + lapatinib, HER2 gene amplification, and the ensuing high levels of HER2 expression on the tumor surface, persist in spite of the tumor progression as determined by HER2 amplified ctDNA levels measured at progression and HER2 IHC findings on rebiopsies of resistant tumors. These findings offer an unexpected 'precision chemotherapy' rescue potential, in spite of progression under anti HER2 treatment and were confirmed experimentally in a HER2 amplified mCRC PDX (metastatic ColoRectal Carcinoma Patient Derived Xenografts), model generated from the viable biopsy of a relapsing HERACLES patient. In this model a randomized trial comparing TDM1 to pertuzumab versus control (6 animal per arm), showed that T-DM1, but not pertuzumab treated animals achieved tumor disappearance. The results of this experiment confirm the principle strength of targeted toxins which is based on their bipartite structure, with one component binding to a disease-specific cell-surface target molecule and the other conferring cytotoxicity, once internalized. In this case HER2 amplification confer to the tumor the characteristics of a 'molecular sponge' for TDM1 with the trastuzumab moiety targeting the still over-abundant HER2 bound to the cell-surface of anti HER2 resistant tumor cell clusters, thus allowing for a 'surgical' delivery of the emtansine cytotoxicity moiety. Given the good predictability of mCRC PDXs model, as testified by HERACLES TRIAL results (NCT03225937), investigators believe that this activity signal should be tested in the clinic. It is therefore proposed a proof-of-concept trial of T-DM1 in HER2 amplified mCRC patients progressing or relapsing after trastuzumab-lapatinib treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histological/confirmed adenocarcinoma of the colon or rectum with metastatic disease not amenable to salvage surgery.
2. Progression (PD) during or after therapy with anti-HER2 therapy including those in HERACLES trial cohort A (trastuzumab and lapatinib) within the HERACLES - A trial.
3. ECOG PS < 2
4. Measurable disease as defined by RECIST 1.1 criteria
5. Adequate hematological function as defined by: ANC >= 1.5 x 10^9/L, platelet count >=100 x 10^9/L, hemoglobin >= 10 g/dL.
6. Adequate renal function, as defined by: creatinine >= 1.5 x UNL
7. Adequate hepatobiliary function, as defined by the following baseline liver function tests:

   1. total serum bilirubin >=1.5 upper normal limit (UNL) (unless documented Gilbert's syndrome )
   2. alanine aminotransferase (ALT), aspartate aminotransferase (AST) >= 2.5xUNL
   3. alkaline phosphatase (AP) >= 2.5xUNL; if total alkaline phosphatase (AP) > 2.5xUNL, alkaline phosphatase liver fraction must be >= 2.5xUNL
8. Adequate contraception for all fertile patients
9. Negative pregnancy test.

Exclusion Criteria:

1. Symptomatic brain metastases
2. Active infection
3. Interval from last anti HER2 therapy < 2 weeks. Patients in treatment with T-DM1 (provided by third-parties) may be eligible for immediate treatment if not in progression at the time of protocol entry.
4. Prior chemotherapy <4 weeks.
5. Impaired cardiac function including any of the following: uncontrolled hypertension (systolic >150 mmHg and/or diastolic > 100 mmHg) or clinically significant (i.e. active) cardiovascular disease: cerebrovascular accident/stroke or myocardial infarction within 6 months prior to first study medication; unstable angina; chronic heart failure (CHF) of New York Heart Association (NYHA) Grade II or higher; or serious cardiac arrhythmia requiring medication, baseline Left Ventricular Ejection Fraction (LVEF) ≤ 55% measured by echocardiography (ECHO)
6. Major surgery in the two weeks prior to entering the clinical trial
7. Concurrent treatment with any other anti-cancer therapy
8. Patient unable to comply with the study protocol owing to psychological, social or geographical reasons
9. Pregnant and lactating women
10. Men and women of childbearing potential who are not using an effective method of contraception
11. Participation in another clinical trial
12. Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2015-07-08 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate according to RECIST 1.1 criteria | every 9 weeks from date of enrollment until the date of first documented progression or date of death for any cause, whichever came first, assessed up to 48 months

SECONDARY OUTCOMES:
Description of the frequency and severity of Adverse Events based on the NCI -CTCAE V4.0 | every 21 days from date of enrollment until the date of first documented progression or date of death for any cause, whichever came first, assessed up to 48 months
Progression Free Survival | every 9 weeks from date of enrollment until the date of first documented progression or date of death for any cause, whichever came first, assessed up to 48 months
  Progression Free Survival

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Fondazione del Piemonte per l'Oncologia, Candiolo
  - Grande Ospedale Metropolitano Niguarda, Milan
  - IOV - Istituto Oncologico Veneto, Padua

IPD SHARING:
Plan to Share IPD: No